CLINICAL TRIAL: NCT04945772
Title: A Phase 2b Randomized, Double-Masked, Sham-Controlled, Study to Evaluate the Efficacy and Safety of Intravitreal Injection of MCO-010 Optogenetic Therapy in Adults With Retinitis Pigmentosa [RESTORE]
Brief Title: Efficacy and Safety of MCO-010 Optogenetic Therapy in Adults With Retinitis Pigmentosa [RESTORE]
Acronym: RESTORE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nanoscope Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: NTXMCO-002.
Record Dates: First submitted 2021-06-15; First posted 2021-06-30 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Retinitis Pigmentosa; Retinitis; Retinal Diseases; Eye Diseases; Eye Diseases, Hereditary; Retinal Dystrophies; Retinal Degeneration
Keywords: Retinitis Pigmentosa; Eye Diseases Hereditary; Eye Diseases; Retinal Degeneration; Inherited Retinal Diseases; Rod & cone dystrophies; Optogenetics; Gene Therapy; AAV vectors; Intravitreal Injections; Low Vision; Multi-Characteristic Opsin; No Light Perception; Visual Acuity; Multi-Luminance Y Mobility Test (MLYMT); Multi-Luminance Shape Discrimination Test (MLSDT)
MeSH Terms: conditions — Retinitis Pigmentosa; Retinitis; Retinal Diseases; Eye Diseases; Eye Diseases, Hereditary; Retinal Dystrophies; Retinal Degeneration; Cone-Rod Dystrophies; Vision, Low | interventions — salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Following a 1:1:1 block randomization schema, 9 subjects will be enrolled in each MCO-010 treatment group, and 9 subjects will be enrolled in the sham-controlled group.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Treatment assignment will be unknown (or masked) to the study participants, the evaluating physician (non-injecting), outcomes assessor, the sponsor and its agents.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- MCO-010- High Dose (Experimental): Participants receive 1.2E11gc/eye of MCO-010
  Interventions: Biological: Gene Therapy Product-MCO-010
- MCO-010- Low Dose (Experimental): Participants receive 0.9E11gc/eye of MCO-010
  Interventions: Biological: Gene Therapy Product-MCO-010
- Sham Injection (Sham Comparator): Participants receive sham injection
  Interventions: Procedure: Sham Injection

INTERVENTIONS:
Biological: Gene Therapy Product-MCO-010 — The MCO-010 is an adeno-associated virus serotype 2-based vector carried multi-characteristic opsin (MCO) gene expression cassette
  Arms: MCO-010- High Dose; MCO-010- Low Dose
Procedure: Sham Injection — Sham Injection
  Arms: Sham Injection

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of a single intravitreal injection of virally-carried Multi-Characteristic Opsin (MCO-010).

DETAILED DESCRIPTION:
This multicenter, randomized, double-masked, sham-controlled, dose-ranging study will evaluate 2 dose levels of MCO-010 in up to 18 subjects with retinitis pigmentosa (9 per dose). An additional nine subjects will receive sham injection. Subjects with a confirmed diagnosis of Advanced Retinitis Pigmentosa (RP) based on clinical examination, dilated fundus examination, and genetic testing will be considered for participation in this study. All subjects will continue to be assessed for 100 weeks following treatment with MCO-010.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Able to comprehend and give informed consent.
3. Confirmed diagnosis of Advanced Retinitis Pigmentosa (RP) based on clinical examination, dilated fundus examination, and genetic testing.
4. Best-Corrected (Freiburg) Visual Acuity worse than 1.9 LogMAR (Snellen equivalent 20/1600) in the study eye and no better than 1.6 LogMAR (Snellen equivalent 20/800) in the fellow eye during screening.

Exclusion Criteria:

Subjects are excluded from the study if any of the following criteria apply:

1. Prior participation in gene therapy program
2. Pre-existing conditions in the study eye such as glaucoma, diseases affecting the optic nerve causing significant visual field loss, active uveitis, corneal or lenticular opacities).
3. Presence of any complicating systemic diseases such as malignancies whose treatment could affect central nervous system function.
4. Active ocular inflammation or recurrent history of idiopathic or autoimmune associated uveitis.
5. Having received retinal prothesis (such as ARGUS-II) or any gene or stem cell therapy (ocular or non-ocular).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-07-13 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2024-01-18 (Actual)

PRIMARY OUTCOMES:
Efficacy of a single intravitreal injection of Multi-Characteristic Opsin (MCO-010) as assessed by best corrected visual acuity. | Week 52
  Change from Baseline in the Freiburg Visual Acuity (quantitative LogMAR) score for the study eye at Week 52.

SECONDARY OUTCOMES:
Efficacy of MCO-010 as assessed by best corrected visual acuity. | Week 76
  Change from Baseline in the Freiburg Visual Acuity (quantitative LogMAR) score for the study eye at Week 76.
Efficacy of MCO-010 as assessed by mobility testing. | Weeks 16,24,32,52,76,100
  Change from Baseline in Multi-Luminance Y-Mobility Test score. Range: -1 to 5, higher score means better outcome.
Efficacy of MCO-010 as assessed by mobility testing. | Weeks 16,24,32,52,76,100
  Proportion of subjects with Multi-Luminance Y-Mobility Test score scores of 2 or more light level improvement from Baseline. Range: 0% to100%, higher score means better outcome.
Efficacy of MCO-010 as assessed by static shape recognition assay. | Weeks 16,24,32,52,76,100
  Proportion of subjects with Multi-Luminance Shape Discrimination Test scores of 2 or more light level improvements from Baseline. Range: 0% to 100%, higher score means better outcome.
Efficacy of MCO-010 as assessed by static shape recognition assay. | Weeks 16,24,32,52,76,100
  Change from Baseline in Multi-Luminance Shape Discrimination Test score. Range: 0 to 5, higher score means better outcome.
Efficacy of MCO-010 as assessed on visual field. | Weeks 16,24,32,52,76,100
  Change from Baseline in Visual Fields measured by Humphrey 30-2 perimetry.

OTHER OUTCOMES:
Efficacy of MCO-010 as assessed by a composite of functional assessments. | Week 52
  Proportion of subjects demonstrating a ≥2 unit improvement from Baseline in EITHER the MLYMT OR the MLSDT score at Week 52.
Safety of MCO-010. | 100 weeks
  Incidences, nature, and severity of ocular and non-ocular treatment emergent adverse events (TEAEs).

CONTACTS AND LOCATIONS:
Overall Officials: Dr Samarendra Mohanty, Study Chair — Nanoscope Therapeutics Inc.
Locations (6):
- United States (5):
  - Nanoscope Clinical Site, Beverly Hills, California
  - Nanoscope Clinical Site, Pensacola, Florida
  - Nanoscope Clinical Site, Fargo, North Dakota
  - Nanoscope Clinical Site, Houston, Texas
  - Nanoscope Clinical Site, McAllen, Texas
- Nanoscope Clinical Site, Arecibo, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
The results of the clinical trial will be made available when the study is completed. The results will be published on this site and be available to conference presentations and publications.
Time Frame: 12 months after the study is completed
Access Criteria: Efficacy and Safety Results